CLINICAL TRIAL: NCT03846128
Title: Impact of Sunitinib Bioavailability on Toxicity and Treatment Efficacy in Patients Treated for Metastatic Renal Cancer
Acronym: BIOSUNTOX
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Other Study IDs: 2017/181/HP
Record Dates: First submitted 2019-01-31; First posted 2019-02-19 (Actual); Last update posted 2019-07-23 (Actual); Status verified 2019-07

CONDITIONS: Metastatic Kidney Cancer
MeSH Terms: conditions — Kidney Neoplasms | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Biological: blood sample — blood sample performed on C1D1, C1D14, C2D1, C3D1 and C6D1

SUMMARY:
Patients treated on the first line of Sunitinib-targeted therapy for metastatic kidney cancer.

Collection of additional blood tubes during routine blood tests for patient follow-up, to evaluate the plasma concentration of Sunitinib and its active metabolite desethyl-Sunitinib (DES)

ELIGIBILITY:
Inclusion Criteria:

* Patient at least 18 years old
* Patient who read and understood the newsletter and signed the consent form
* Renal cell carcinoma histologically proven stage IV
* Metastatic stage proven on CT, synchronous or metachronous examination
* Patient operated on or not from the primary tumor
* Eligible for first-line systemic therapy with Sunitinib-targeted therapy for oncology urology
* Affiliation to a social security scheme
* Effective contraception (as defined by the WHO) for at least 3 months at the inclusion visit, during treatment and for 1 month after the end of the research (negative pregnancy test)
* Postmenopausal woman: confirmatory diagnosis (amenorrhea not clinically induced for more than 12 months at inclusion visit)
* General condition WHO 0 to 2
* Life expectancy estimated at more than 6 months at baseline

Exclusion Criteria:

* Non-metastatic disease
* Other cancer proven histologically, or in complete remission for less than 2 years
* Contraindication to SUTENT 50 mg hard capsules: Hypersensitivity to the active substance or to any of the excipients
* History of immunotherapy treatment for kidney cancer, previous treatment with targeted therapies for the same or previous cancer
* Pregnant or lactating woman or wishing to breastfeed within 6 months after the last treatment or no known contraception,
* Person deprived of liberty by an administrative or judicial decision or person placed under the protection of justice / sub-guardianship or curatorship
* Patient currently involved in an interventional trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients treated on the first line of Sunitinib-targeted therapy for metastatic kidney cancer
Sampling Method: Probability Sample
Enrollment: 64 (Estimated)
Dates: Start 2019-08 (Estimated); Primary Completion 2024-05 (Estimated); Study Completion 2024-05 (Estimated)

PRIMARY OUTCOMES:
hazard ratio of a severe toxicity, grade 3-4 clinical and / or biologicalas according to the plasma concentration of Sunitinib | At the end of Cycle 1 (each cycle is 28 days)
  hazard ratio of a severe toxicity, grade 3-4 clinical and / or biologicalas according to the plasma concentration of Sunitinib
hazard ratio of a severe toxicity, grade 3-4 clinical and / or biologicalas according to the plasma concentration of Sunitinib | At the end of Cycle 2 (each cycle is 28 days)
  hazard ratio of a severe toxicity, grade 3-4 clinical and / or biologicalas according to the plasma concentration of Sunitinib
hazard ratio of a severe toxicity, grade 3-4 clinical and / or biologicalas according to the plasma concentration of Sunitinib | At the end of Cycle 3 (each cycle is 28 days)
  hazard ratio of a severe toxicity, grade 3-4 clinical and / or biologicalas according to the plasma concentration of Sunitinib
hazard ratio of a severe toxicity, grade 3-4 clinical and / or biologicalas according to the plasma concentration of Sunitinib | At the end of Cycle 4 (each cycle is 28 days)
  hazard ratio of a severe toxicity, grade 3-4 clinical and / or biologicalas according to the plasma concentration of Sunitinib
hazard ratio of a severe toxicity, grade 3-4 clinical and / or biologicalas according to the plasma concentration of Sunitinib | At the end of Cycle 5 (each cycle is 28 days)
  hazard ratio of a severe toxicity, grade 3-4 clinical and / or biologicalas according to the plasma concentration of Sunitinib
hazard ratio of a severe toxicity, grade 3-4 clinical and / or biologicalas according to the plasma concentration of Sunitinib | At the end of Cycle 6 (each cycle is 28 days)
  hazard ratio of a severe toxicity, grade 3-4 clinical and / or biologicalas according to the plasma concentration of Sunitinib
hazard ratio of a severe toxicity, grade 3-4 clinical and / or biological according to the plasma concentration of desethyl-Sunitinib | At the end of Cycle 1 (each cycle is 28 days)
  hazard ratio of a severe toxicity, grade 3-4 clinical and / or biological according to the plasma concentration of desethyl-Sunitinib
hazard ratio of a severe toxicity, grade 3-4 clinical and / or biological according to the plasma concentration of desethyl-Sunitinib | At the end of Cycle 2 (each cycle is 28 days)
  hazard ratio of a severe toxicity, grade 3-4 clinical and / or biological according to the plasma concentration of desethyl-Sunitinib
hazard ratio of a severe toxicity, grade 3-4 clinical and / or biological according to the plasma concentration of desethyl-Sunitinib | At the end of Cycle 3 (each cycle is 28 days)
  hazard ratio of a severe toxicity, grade 3-4 clinical and / or biological according to the plasma concentration of desethyl-Sunitinib
hazard ratio of a severe toxicity, grade 3-4 clinical and / or biological according to the plasma concentration of desethyl-Sunitinib | At the end of Cycle 4 (each cycle is 28 days)
  hazard ratio of a severe toxicity, grade 3-4 clinical and / or biological according to the plasma concentration of desethyl-Sunitinib
hazard ratio of a severe toxicity, grade 3-4 clinical and / or biological according to the plasma concentration of desethyl-Sunitinib | At the end of Cycle 5 (each cycle is 28 days)
  hazard ratio of a severe toxicity, grade 3-4 clinical and / or biological according to the plasma concentration of desethyl-Sunitinib
hazard ratio of a severe toxicity, grade 3-4 clinical and / or biological according to the plasma concentration of desethyl-Sunitinib | At the end of Cycle 6 (each cycle is 28 days)
  hazard ratio of a severe toxicity, grade 3-4 clinical and / or biological according to the plasma concentration of desethyl-Sunitinib

SECONDARY OUTCOMES:
plasma desethyl-Sunitinib (DES) concentration | Cycle1 Day14 (each cycle is 28 days)
  influence of plasma DES concentration on patients survival
plasma Sunitinib concentration | Cycle1 Day14 (each cycle is 28 days)
  influence of plasma Sunitinib concentration on patients survival
plasma Sunitinib concentration | Cycle1 Day28 (each cycle is 28 days)
  influence of plasma Sunitinib concentration on patients survivall
plasma DES concentration | Cycle1 Day28 (each cycle is 28 days)
  influence of plasma Sunitinib concentration on patients survival
plasma Sunitinib concentration | Cycle2 Day28(each cycle is 28 days)
  influence of plasma Sunitinib concentration on patients survival
plasma DES concentration | Cycle2 Day28 (each cycle is 28 days)
  influence of plasma DES concentration on patients survival
plasma Sunitinib concentration | Cycle3 Day28 (each cycle is 28 days)
  influence of plasma Sunitinib concentration on patients survival
plasma DES concentration | Cycle3 Day28 (each cycle is 28 days)
  Evaluate the influence of plasma DES concentration on patients survival
plasma Sunitinib concentration | Cycle6 Day28 (each cycle is 28 days)
  influence of plasma Sunitinib concentration on patients survival
plasma DES concentration | Cycle6 Day28 (each cycle is 28 days)
  influence of plasma DES concentration on patients survival